CLINICAL TRIAL: NCT00361387
Title: Randomized, Double-Blind, Placebo-Controlled Study of Dexmethylphenidate Hydrochloride, (d-MPH) in the Treatment of Fatigue in Sarcoidosis Subjects.
Brief Title: Use of Focalin for Fatigue in Sarcoidosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Robert P. Baughman MD, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-02-23-03
Record Dates: First submitted 2006-08-07; First posted 2006-08-08 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Sarcoidosis
Keywords: Sarcoidosis; Sarcoid
MeSH Terms: conditions — Sarcoidosis | interventions — Methylphenidate; Dexmethylphenidate Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: d-methylphenidate — oral dosing for 8 weeks then cross over to placebo in random order
  Other Names: Focalin

SUMMARY:
Patients diagnosed with chronic sarcoidosis with fatigue for more than 6 months. Sarcoidosis and its treatment can greatly affect your quality of life. Many patients suffer from fatigue (feeling tired), lack of focus and concentration, in ability to organize their daily activities, and memory loss. These commonly reported symptoms often get in the way of everyday life.

DETAILED DESCRIPTION:
This is to be a double blind, randomized trial with cross over of 12 patients with chronic sarcoidosis on stable systemic therapy. Patients will be screened for fatigue using a modified SNAP and Facit-F scores. Patients will be in the study for 20 weeks. Objective of study: To determine the effect of dexmethylphenidate hydrochloride, (d-MPH)(Focalin) on fatigue in Sarcoidosis. The is a common complaint in sarcoidosis, related to the chronic inflammatory nature of the disease. It may also related to therapy for the disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sarcoidosis using standard criteria
* Disease for more than one year
* Complain of fatigue which has been present for more than six months.
* Over 18 years of age

Exclusion Criteria:

* Pregnancy
* Change in therapy for sarcoidosis in prior three months
* history of ventricular arrythmias
* Patients with a history of anxiety disorder, glaucoma, motor ties or a family history of Tourette's syndrome.
* Patients who are currently receiving or have received monoamine oxidase inhibitors within 14 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Improvement of fatigue. | 30 weeks

SECONDARY OUTCOMES:
Improvement of pulmonary status | 30 weeks
Safety of treatment | 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Baughman, MD, Principal Investigator — Unversity of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Lower EE, Harman S, Baughman RP. Double-blind, randomized trial of dexmethylphenidate hydrochloride for the treatment of sarcoidosis-associated fatigue. Chest. 2008 May;133(5):1189-95. doi: 10.1378/chest.07-2952. Epub 2008 Feb 8. PMID 18263672